CLINICAL TRIAL: NCT01384032
Title: Apolipoprotein E Genotype as a Determinant of LDL-cholesterol Response to Dietary Fat Manipulation
Brief Title: Study Into Genetic Influence on Cholesterol Response to Dietary Fat
Acronym: Satgene
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Reading (Other)
Collaborators: Wellcome Trust (Other)
Responsible Party: Professor Julie Lovegrove, Department of Food and Nutritional Sciences, University of Reading
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: WT085045MA
Record Dates: First submitted 2011-06-20; First posted 2011-06-28 (Estimated); Last update posted 2011-06-28 (Estimated); Status verified 2011-06

CONDITIONS: Cardiovascular Diseases
Keywords: CVD, LDL-C, apoE, SFA, DHA
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Diet, Fat-Restricted

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Low fat diet (Experimental): Subjects were asked to consume a low fat diet for 8 weeks. Composition: 28% energy from fat, 8% energy from saturated fat, 55% energy from carbohydrate. Subjects were provided with low fat spread, cooking oil and snacks and asked to consume these in place of normally eaten equivalent foods. Subjects were asked to consume two extra portions of carbohydrate per day (e.g. two slices of bread, equivalent to 35g carbohydrate) and to consume low fat dairy products. Subjects also consumed 2g control oil per day during this period. Control oil comprised palm olein and soybean oil.
  Interventions: Dietary Supplement: Low fat diet
- High saturated fat diet (Experimental): Subjects were asked to consume a high saturated fat diet for 8 weeks. Composition: 38% energy from fat, 18% energy from saturated fat, 45% energy from carbohydrate. Subjects were provided with spread, cooking oil and snacks and asked to consume these in place of normally eaten equivalent foods. Subjects were asked to consume one less portion of carbohydrate per day (e.g. one slice of bread and to consume full fat dairy products. Subjects also consumed 2g control oil per day during this period. Control oil comprised palm olein and soybean oil.
  Interventions: Dietary Supplement: Hgih saturated fat diet
- High saturated fat plus DHA diet (Experimental): Subjects were asked to consume a high saturated fat diet for 8 weeks. Composition: 38% energy from fat, 18% energy from saturated fat, 45% energy from carbohydrate. Subjects were provided with spread, cooking oil and snacks and asked to consume these in place of normally eaten equivalent foods. Subjects were asked to consume one less portion of carbohydrate per day (e.g. one slice of bread and to consume full fat dairy products. Subjects also consumed 6g DHA-rich oil per day during this period providing 3g DHA.
  Interventions: Dietary Supplement: High saturated fat diet

INTERVENTIONS:
Dietary Supplement: Low fat diet — Subjects were asked to consume a low fat diet for 8 weeks. Composition: 28% energy from fat, 8% energy from saturated fat, 55% energy from carbohydrate. Subjects were provided with low fat spread, cooking oil and snacks and asked to consume these in place of normally eaten equivalent foods. Subjects were asked to consume two extra portions of carbohydrate per day (e.g. two slices of bread, equivalent to 35g carbohydrate) and to consume low fat dairy products. Subjects also consumed 2g control oil per day during this period. Control oil comprised palm olein and soybean oil.
  Arms: Low fat diet
Dietary Supplement: Hgih saturated fat diet — Subjects were asked to consume a high saturated fat diet for 8 weeks. Composition: 38% energy from fat, 18% energy from saturated fat, 45% energy from carbohydrate. Subjects were provided with spread, cooking oil and snacks and asked to consume these in place of normally eaten equivalent foods. Subjects were asked to consume one less portion of carbohydrate per day (e.g. one slice of bread and to consume full fat dairy products. Subjects also consumed 2g control oil per day during this period. Control oil comprised palm olein and soybean oil.
  Arms: High saturated fat diet
Dietary Supplement: High saturated fat diet — Subjects were asked to consume a high saturated fat diet for 8 weeks. Composition: 38% energy from fat, 18% energy from saturated fat, 45% energy from carbohydrate. Subjects were provided with spread, cooking oil and snacks and asked to consume these in place of normally eaten equivalent foods. Subjects were asked to consume one less portion of carbohydrate per day (e.g. one slice of bread and to consume full fat dairy products. Subjects also consumed 6g DHA-rich oil per day during this period providing 3g DHA.
  Arms: High saturated fat plus DHA diet

SUMMARY:
Cardiovascular disease (CVD) is recognised as one of the main causes of death in the western world. LDL- cholesterol ('bad' cholesterol) and other lipids (fats) are important CVD risk factors. Apolipoprotein E (apoE) is an important transporter of fats in the blood. ApoE comes in E2, E3 and E4 forms, depending on your genetic make up. Approximately 60% of the UK population are E3/E3, 25% E4 carriers and 15% E2 carriers. There is some evidence to suggest that an E4 genotype may put you at modestly higher risk of CVD. Furthermore although very inconclusive previous studies have suggested that E4 individuals are slightly more sensitive to the LDL-cholesterol modifying effects of dietary fats (saturated fat, total fat, fish oil) showing slightly, greater reductions when low levels of these fat are consumed, and greater increases when high levels of these fat are consumed. Therefore, the aims of the Satgene study is to examine the impact of modifications in dietary total fat and saturated fat intakes, alone and in combination with fish oil supplement on LDL-cholesterol and other blood lipids, in individuals with an E3 and E4 genotype. The levels of total fat and saturated fat used in the current study are within the range observed in a typical UK population.

ELIGIBILITY:
Inclusion Criteria:

Men & women 35-70 years BMI 20-32 kg/m2 Haemoglobin (anaemia): 12.5-18.0g/l (men) and > 11.5-16g/l (women) Gamma GT (liver function) (< 80 IU/l), Triglyceride (between 1-4 mmol/l), Plasma total cholesterol (4.5-8 mmol/l) Glucose (World Health organisation recommend <7 mmol/L).

Exclusion Criteria:

* Females who are breast feeding, may be pregnant, or if child-bearing potential are not taking effective contraceptive precautions
* Likely to alter oral contraceptive or HRT usage during the course of the study
* Blood Pressure > 160/100 mm Hg (UK guidelines for stage 2 hypertension)
* Had suffered a myocardial infarction or stroke in the previous 12 months
* Hypertensive medication
* Diabetics type I and II
* Any volunteers on a weight reducing diet, or vegan/vegetarians as study requires consumption of dairy products and fish oils
* On high dose fish oil supplements (> 1g EPA + DHA per day)
* Elevated lipids requiring medication such as statins, fibrates, gall bladder problems or other abnormalities of fat metabolism
* Subjects not willing to make the necessary dietary changes during the study
* Subjects drinking excessive alcohol (UK recommendations/wk currently for men are, no more than 21 units of alcohol per week or more than four units in any one day. For women, no more than 14 units of alcohol per week or more than three units per day).
* Subjects who train at a high level, or attend more than 3 hours organised exercise classes per week

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2009-01; Primary Completion 2010-10 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Change in low density lipoprotein cholesterol (LDL-C) | 0, 8, 16, and 24 weeks

SECONDARY OUTCOMES:
Change in arterial stiffness | 0, 8, 16, 24 weeks
  Arterial stiffness is a measure of vascular reactivity. This was assessed by Digital Volume Pulse using Pulse Trace PCA2 Machine (Micromedical, UK)
Change in fasting glucose | 0, 8, 16, 24 weeks
Change in fasting insulin | 0, 8, 16, 24 weeks
Change in fasting triglycerides (TAG) | 0, 8, 16, 24 weeks
Change in C-reactive protein (CRP) | 0, 8, 16, 24 weeks
Change in blood pressure | 0, 8, 16, 24 weeks
Change in body weight | 0, 8, 16, 24 weeks
Change in plasma phospholipid fatty acids | 0, 8, 16, 24 weeks
Change in total cholesterol | 0, 8, 16, 24 weeks
Change in high-density lipoprotein cholesterol (HDL) | 0, 8, 16, 24 weeks
Change in apolipoproteins B, CIII and E | 0, 8, 16, 24 weeks
Change in very low density lipoprotein (VLDL) | 0, 8, 16, 24 weeks
Change in chylomicrons (CM) | 0, 8, 16, 24 weeks
Change in inflammatory cytokine production | 9, 8, 16, 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Julie A Lovegrove, Professor, Principal Investigator — University of Reading
Locations (1):
- Department of Food and Nutritional Sciences, University of Reading, Reading, United Kingdom

REFERENCES:
- [Derived] Chouinard-Watkins R, Conway V, Minihane AM, Jackson KG, Lovegrove JA, Plourde M. Interaction between BMI and APOE genotype is associated with changes in the plasma long-chain-PUFA response to a fish-oil supplement in healthy participants. Am J Clin Nutr. 2015 Aug;102(2):505-13. doi: 10.3945/ajcn.114.103507. Epub 2015 Jun 17. PMID 26085515
- [Derived] Carvalho-Wells AL, Jackson KG, Lockyer S, Lovegrove JA, Minihane AM. APOE genotype influences triglyceride and C-reactive protein responses to altered dietary fat intake in UK adults. Am J Clin Nutr. 2012 Dec;96(6):1447-53. doi: 10.3945/ajcn.112.043240. Epub 2012 Nov 7. PMID 23134888
- [Derived] Lockyer S, Tzanetou M, Carvalho-Wells AL, Jackson KG, Minihane AM, Lovegrove JA. SATgenepsilon dietary model to implement diets of differing fat composition in prospectively genotyped groups (apoE) using commercially available foods. Br J Nutr. 2012 Nov 14;108(9):1705-13. doi: 10.1017/S0007114511007082. Epub 2012 Jan 16. PMID 22243632